CLINICAL TRIAL: NCT04387604
Title: Effect of the Vitreous in Response to Intravitreal (IV) Injections of Ranibizumab (0.5mg/0.05ml) for the Treatment of Diabetic Macular Edema
Brief Title: Effect of the Vitreous in Response to Intravitreal Injections of Ranibizumab for the Treatment of Diabetic Macular Edema
Acronym: DEVITRA
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Bernardete Pessoa MD, Senior Specialist Vitreoretinal Surgeon, Centro Hospitalar do Porto
Other Study IDs: 2017080120190301
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- non vitrectomized eyes: ranibizumab injections (0.5 mg/0.05ml) following a PRN regimen
  Interventions: Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS]
- vitrectomized eyes: ranibizumab injections (0.5 mg/0.05ml) following a PRN regimen
  Interventions: Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS]

INTERVENTIONS:
Drug: Ranibizumab 0.5 MG/0.05 ML Intraocular Solution [LUCENTIS] — PRN regimen. Treatment Schedule Repeat injections at every 4-week visit if eye "improves" or "worsens" (defined as ≥5 letter change from last injection or ≥10% CST change on OCT from last injection or CSF>300 μm at any timepoint).
  Defer injections if either BCVA of 85 letters and OCT CSF "normal" (CSF≤300 μm and non-existent intra- or sub-retinal fluid); or OCT CSF "normal" (CSF≤300 μm) and stable BCVA (defined as < 5 letters change from last injection) after two consecutive injections during the first 24 weeks, or after one injection if the initial stability period has already been achieved (OCT CSF "normal" and stable BCVA).
  Resume injections if BCVA or OCT worsens.

SUMMARY:
PURPOSE: To evaluate the effect of the vitreous in response to intravitreal (IV) injections of ranibizumab 0.5 mg/0.05ml (Lucentis; Genentech, South San Francisco, CA) for the treatment of diabetic macular edema (DME).

METHODS: Prospective, observational, multicenter study, conducted at Centro Hospitalar e Universitário do Porto, Portugal. Best-corrected visual acuity and central foveal thickness will be evaluated at baseline and every month until the end of follow-up. OCT biomarkers such as retinal layers thickness will also be analyzed.

A p value of 0.05 or less will be considered to be statistically significant. HYPOTHESIS: Vitrectomized patients will improve less than non-vitrectomized patients.

DETAILED DESCRIPTION:
Patients will be included in two different groups according to the vitreous status: group 1 - non vitrectomized eyes; group 2 - vitrectomized eyes. Patients will be followed-up according to the standard of care and a final analysis of the results will be performed at 12+/-1 months of follow-up, which is the minimum follow-up period required for each patient. In group 1 the effect of VMA existence and PVD status will also be analyzed. The recruitment period will be of 6 months.

Treatment All patients will be treated with IV ranibizumab injections (0.5 mg/0.05ml) following a PRN regimen. The injections will be performed in the operating room following the standard intravitreal injections protocol. When required, adjunct treatment, with macular and/or peripheral LASER (rescue LASER), will be also admitted at or after 24 weeks if persistent DME not improving after at least 2 injections.

Treatment Schedule Repeat injections at every 4-week visit if eye "improves" or "worsens" (defined as ≥5 letter change from last injection or ≥10% CST change on OCT from last injection or CSF>300 μm at any timepoint).

Defer injections if either BCVA of 85 letters and OCT CSF "normal" (CSF≤300 μm and non-existent intra- or sub-retinal fluid); or OCT CSF "normal" (CSF≤300 μm) and stable BCVA (defined as < 5 letters change from last injection) after two consecutive injections during the first 24 weeks, or after one injection if the initial stability period has already been achieved (OCT CSF "normal" and stable BCVA).

Resume injections if BCVA or OCT worsens.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age with either type 1 or type 2 diabetes mellitus;
* maximal central subfield foveal thickness (CSF) of at least 300μm (according to SD-OCT images - Spectral Domain Optical Coherence Tomography);
* BCVA of 20 to 80 letters, using ETDRS letters chart;
* ability to provide written informed consent.

Exclusion Criteria:

* Pregnant or lactating;
* Epiretinal membrane (ERM) existence in the study eye;
* persistent posterior hyaloid adherence after vitrectomy for group 2;
* previous vitrectomy for group 1;
* history of other retinal vascular diseases in the study eye;
* LASER photocoagulation or intravitreal injections (IV) of anti-VEGF or systemic anti-VEGF or pro-anti-VEGF treatment and cataract surgery in the 6 months previously to the study eye inclusion;
* IV or peribulbar corticosteroid injections in the 6 months previously to study eye inclusion;
* history of IV of implant of fluocinolone acetonide in the study eye;
* vitreous hemorrhage or opacification in the study eye;
* active proliferative diabetic retinopathy in the study eye;
* active ocular inflammation or infection in either eye;
* aphakia in the study eye;
* other causes for macular edema, for example, after cataract surgery in the study eye;
* other causes of visual loss in the study eye;
* other diseases that may affect the course of macular edema in the study eye;
* uncontrolled glaucoma in either eye (intraocular pressure > 24 mmHg with treatment);
* history of arterial thrombotic event in the previous 6 months;
* uncontrolled arterial hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure > 100 mmHg);
* ward of the state.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with DME followed on the ocular diabetes consultation of Centro Hospitalar e Universitário do Porto, Portugal, or Hospital Santa Maria Maior de Barcelos, Portugal, either non vitrectomized or vitrectomized.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
assess the number of IV injections needed to control DME between groups | 18 months
  DME control is defined as 1) BCVA of 85 letters and OCT CFT "normal" (CFT≤300 μm and non-existent intra- or sub-retinal fluid); or 2) OCT CFT "normal" (CFT≤300 μm) and stable BCVA (defined as <5 letters change from last injection) after two consecutive injections during the first 24 weeks, or after one injection if the initial stability period has already been achieved (OCT CFT "normal" and stable BCVA).

SECONDARY OUTCOMES:
compare the functional changes at the end of follow-up between groups | 18 months
  Functional change will be measured by the Early Treatment Diabetic Retinopathy Scale (ETDRS) which measures the best-corrected visual acuity with an ETDRS-like chart at 4 meters in number letters or at 1 meter when patients are unable to read any letters on the ETDRS chart at 4 meters. The ETDRS scale varies from 1 to 85 letters (85 letters correspond to a 20/20 in the Snellen scale).
  The higher the value the better the outcome. A clinical significant functional improvement will be considered for a gain of ≥5 EDTRS letters.
compare the anatomical changes at the end of follow-up between groups | 18 months
  Anatomical change will be measured by central foveal thickness (CFT), measured by Optical Coherence Tomography, automatically measured by the software in the central 1 mm. A CFT <240µm or >300 µm is considered pathological. A CFT between 240 and 300 µm is considered physiological. CFT has no defined minimum or maximum values.
  Since patients with diabetic macular edema usually have CFT >300 µm the goal of treatment is to lower the CFT to values between 240 and 300 µm. A clinical significant anatomical improvement will be considered for a change in CFT≥10%.
compare the percentage of type of responder during the follow-up period between groups | 18 months
  Type of responder is defined as follows:
  * good responder: when beyond the 24th week of follow-up (maximum 7 injections) there was a complete anatomical response (CFT≤300μm) with an increase in BCVA ≥5 letters;
  * non-responder: 13 injections and final CFT >400 um or ≤10% of CFT reduction and BCVA decrease (or BCVA gain <5 letters)
  * incomplete responder: between good and non-responder criteria.
access the percentage, in group 2, of focal VMA and PVD status and type of response | 18 months
  to access the percentage, in group 2, of focal VMA and PVD status, and if those changed during the follow-up period influenced the type of response
assess retinal layers thickness as prognostic and pathophysiological biomarkers of DME treatment response | 18 months
  * to assess baseline retinal layers thickness correlation with final BCVA
  * to assess the influence of the variation of retinal layers thickness (baseline versus final) on final BCVA
  * to assess differences between groups according to the above points;
  * to associate the type of responder and baseline and final retinal layers thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardete Pessoa, MD, Principal Investigator — Centro Hospitalar e Universitário do Porto
Locations (1):
- Hospital de Santo António, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pessoa B, Leite J, Ferreira A, Ramalhao J, Pocas J, Jose D, Coelho C, Figueira J, Meireles A, Beirao JM. Oct biomarkers for early prognosis in diabetic macular edema treatment with ranibizumab. Eur J Ophthalmol. 2024 Jul;34(4):1141-1148. doi: 10.1177/11206721231210753. Epub 2023 Nov 3. PMID 37919940
- [Derived] Pessoa B, Leite J, Heitor J, Coelho J, Monteiro S, Coelho C, Figueira J, Meireles A, Melo-Beirao JN. Vitrectomized versus non-vitrectomized eyes in diabetic macular edema response to ranibizumab-retinal layers thickness as prognostic biomarkers. Sci Rep. 2021 Nov 29;11(1):23055. doi: 10.1038/s41598-021-02532-4. PMID 34845300
- [Derived] Pessoa B, Marques JH, Leite J, Silva N, Jose D, Coelho C, Figueira J, Meireles A, Melo-Beirao JN. Choroidal Blood Flow After Intravitreal Ranibizumab in Vitrectomized and Non-Vitrectomized Eyes with Diabetic Macular Edema. Clin Ophthalmol. 2021 Oct 9;15:4081-4090. doi: 10.2147/OPTH.S325037. eCollection 2021. PMID 34675476